CLINICAL TRIAL: NCT01438216
Title: Anidulafungin Population Kinetics in the Intensive Care Population
Brief Title: Anidulafungin Pharmacokinetics in Intensive Care Unit Patients
Acronym: ANICK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, V.M. Middel-Baars, PharmD, hospital pharmacist trainee, Amsterdam UMC, location VUmc
Other Study IDs: ANIPKIC001; 2011-001911-30 (EudraCT Number)
Record Dates: First submitted 2011-09-14; First posted 2011-09-22 (Estimated); Last update posted 2011-09-22 (Estimated); Status verified 2011-09

CONDITIONS: Invasive Candidiasis; Candidemia
Keywords: Pharmacokinetics; Intensive Care; Candidemia; Invasive candidiasis; Anidulafungin
MeSH Terms: conditions — Candidiasis, Invasive; Candidemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- VUmc IC: Due to multicentre, 2 groups of patient in 1 cohort
- UMCN IC: Due to multicentre, 2 groups of patient in 1 cohort

SUMMARY:
The purpose of this study is to determine the pharmacokinetics of anidulafungin in intensive care patients.

DETAILED DESCRIPTION:
Not a lot is known about the pharmacokinetic profile of anidulafungin in IC-patients. IC-patients are at high(er) risk for getting a systemic mould/yeast infection. Anidulafungin is a safe echinocandin with, so far, no reported interactions and few adverse effects. Due to this, anidulafungin is used more often on IC-wards. It is part of the national (Netherlands) IC sepsis protocol. The factors that influence the pharmacokinetics of anidulafungin in IC-patients has not been studied yet. Because these factors are unknown for this population, it is necessary for this research to be done.

Any patient with an (suspected) invasive candidiasis whom is treated with anidulafunging can be includen.

20 patients will be included from 2 different university hospital (10 each). Samples will be taken on different days and timepoints, troughlevels on all treatment days and on treatment day 3 and 7 more samples will be taken voor AUC calculations.

ELIGIBILITY:
Inclusion Criteria:

* Patient is admitted to the intensive care unit
* Patient has a central (venous) infusion line
* Patient is at least 18 years old
* Patient receives treatment with anidulafungin

  * that is initiated on the ICU or
  * that is continued on the ICU and the patient has had no more than 2 days of treatment with anidulafungin

Exclusion Criteria:

* Documented history of sensitivity to medicinal products or excipients similar to those found in the anidulafungin preparation
* Patient receives treatment with anidulafungin that is continued on the ICU and the patient has had 3 or more days of treatment with anidulafungin
* A woman that is pregnant, wanting to become pregnant or nursing an infant
* < 48 hours (expected) treatment with anidulafungin on the ICU ward
* Has previously participated in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive Care patients
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-02 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic population model for anidulafungin for the ICU population | 1 year, after inclusion of 20 patients
  The populationmodel will be created with NONMEM. The concentrations in the bloodsamples will be the input source for this model.

SECONDARY OUTCOMES:
Time until clinical and microbiological response is reached | 1 year, after inclusion of 20 patients
  Registration of time till response
To determine the covariates that influence the kinetics of anidulafungin. | 1 year, after inclusion of 20 patients
  With the help from modeling program NONMEM
To determine the optimal dosage(scheme) for intensive care patients. | 1 year, after inclusion of 20 patients
  Calculation of optimal dosage can be done by NONMEM.
To determine which of the two ratios is the most predictive voor clinical outcome: AUC/MIC or Cmax/MIC. | 1 year, after inclusion of 20 patients
  If the actual MIC is known, this can can be determined.
Registration of side effects and adverse events | 1 year, after inclusion of 20 patients
  To register safety od anidulafungin use on ICU

CONTACTS AND LOCATIONS:
Overall Officials: Vera M Middel-Baars, PharmD, Principal Investigator — Amsterdam UMC, location VUmc; Eleonora L Swart, PhD, Principal Investigator — Amsterdam UMC, location VUmc; Roger Brüggemann, PharmD, Principal Investigator — Radboud University Nijmegen Medical Center
Locations (2):
- Netherlands (2):
  - Radboud University Nijmegen Medical Center, Nijmegen, Gelderland
  - VU University Medical Center, Amsterdam, North Holland

REFERENCES:
- [Derived] Bruggemann RJ, Middel-Baars V, de Lange DW, Colbers A, Girbes AR, Pickkers P, Swart EL. Pharmacokinetics of Anidulafungin in Critically Ill Intensive Care Unit Patients with Suspected or Proven Invasive Fungal Infections. Antimicrob Agents Chemother. 2017 Jan 24;61(2):e01894-16. doi: 10.1128/AAC.01894-16. Print 2017 Feb. PMID 27872072